CLINICAL TRIAL: NCT03550794
Title: Thiamine as a Renal Protective Agent in Septic Shock: A Randomized, Controlled Study
Brief Title: Thiamine as a Renal Protective Agent in Septic Shock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Michael Donnino, Associate Professor of Emergency Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018P-000204
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Sepsis; Kidney Injury; Thiamine Deficiency
MeSH Terms: conditions — Sepsis; Thiamine Deficiency | interventions — thiamine hydrochloride; Thiamine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A randomization list will be prepared by an independent statistician using 1:1 randomization in blocks of two and four. This list will be provided to the research pharmacy, and the research pharmacy will be the only unblinded people involved with the study, and will have no patient contact or role in the analysis or other aspects of the study. Thiamine is colorless and odorless, and the 200mg dose is mixed in 5mL of normal saline. Placebo will be 50mL of normal saline and is indistinguishable in appearance from thiamine. Study team, clinical team and patient and family will all be blind to the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Thiamine (Experimental): 200mg parenterally administered thiamine hydrochloride given twice daily for a 3 days (6 doses)
  Interventions: Drug: Thiamine Hydrochloride
- Placebo (Placebo Comparator): Matching placebo (50ml 0.9%NACL) given twice daily for 3 days (6 administrations)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Thiamine Hydrochloride — Thiamine hydrochloride is a water soluble vitamin (vitamin B1). 200mg of thiamine hydrochloride in 50ml 0.9%NACL will be administered twice daily for 3 days.
  Other Names: Thiamine; Vitamin B1
  Arms: Thiamine
Drug: Placebo — 50ml of 0.9% NACL will serve as the placebo
  Other Names: Normal Saline; 0.9%NACL
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo controlled study to investigate the effect of intravenous thiamine (vitamin B1) on renal function in septic shock.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled study to investigate the effect of intravenous thiamine (vitamin B1) on renal injury in septic shock. Patients admitted with septic shock who have a lactate of at least 2.0mmol/L and do not have pre-existing renal failure requiring dialysis will be eligible for the study. Enrolled patients will be randomized to intravenous thiamine 200mg twice daily for 6 doses or matching placebo. Blood will be drawn at several time points to assess biomarkers of renal injury. Secondary endpoints include need for renal replacement therapy, length of ICU stay, and hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥18 years of age
2. Suspected or Confirmed Infection (defined as collection of a blood/fluid culture and provision of an antimicrobial)
3. Receipt of a vasopressor agent (e.g. norepinephrine, phenylephrine, vasopressin)
4. Serum lactate ≥2mmol/L
5. Creatinine >1.0mg/dL

Exclusion Criteria:

1. Clinical indication for thiamine administration (alcoholism, known or highly suspected deficiency) or treatment with thiamine beyond the amount found in a standard multivitamin within the last 10 days
2. Renal replacement therapy within the past 30 days
3. Comfort measures only or anticipated withdrawal of support within 24 hours
4. Protected populations (pregnant women, prisoners)
5. Known thiamine allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ari Moskowitz, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (4):
- United States (4):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Northshore University Hospital, Manhasset, New York
  - Montefiore Medical Center, New York, New York
  - Long Island Jewish Hospital, Queens, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Moskowitz A, Andersen LW, Cocchi MN, Karlsson M, Patel PV, Donnino MW. Thiamine as a Renal Protective Agent in Septic Shock. A Secondary Analysis of a Randomized, Double-Blind, Placebo-controlled Trial. Ann Am Thorac Soc. 2017 May;14(5):737-741. doi: 10.1513/AnnalsATS.201608-656BC. PMID 28207287
- [Background] Donnino MW, Andersen LW, Chase M, Berg KM, Tidswell M, Giberson T, Wolfe R, Moskowitz A, Smithline H, Ngo L, Cocchi MN; Center for Resuscitation Science Research Group. Randomized, Double-Blind, Placebo-Controlled Trial of Thiamine as a Metabolic Resuscitator in Septic Shock: A Pilot Study. Crit Care Med. 2016 Feb;44(2):360-7. doi: 10.1097/CCM.0000000000001572. PMID 26771781
- [Derived] Vine J, Lee JH, Kravitz MS, Grossestreuer AV, Balaji L, Leland SB, Berlin N, Moskowitz A, Donnino MW. Thiamine administration in septic shock: a post hoc analysis of two randomized trials. Crit Care. 2024 Feb 6;28(1):41. doi: 10.1186/s13054-024-04818-1. PMID 38321529
- [Derived] Moskowitz A, Berg KM, Grossestreuer AV, Balaji L, Liu X, Cocchi MN, Chase M, Gong MN, Gong J, Parikh SM, Ngo L, Berlin N, Donnino MW. Thiamine for Renal Protection in Septic Shock (TRPSS): A Randomized, Placebo-controlled, Clinical Trial. Am J Respir Crit Care Med. 2023 Sep 1;208(5):570-578. doi: 10.1164/rccm.202301-0034OC. PMID 37364280

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Thiamine | Placebo
Started | 46 | 49
Completed | 42 | 46
Not Completed | 4 | 3
Not completed — No longer met inclusion criteria | 1 | 2
Not completed — Goals of care changed | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thiamine | Placebo | Total
Number analyzed (Participants) | 42 | 46 | 88
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 74.5 [64.0 to 83.8] | 70.0 [61.0 to 78.0] | 71.5 [61.0 to 81.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 19 | 43
  Male | 18 | 27 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Native Alaskan | 0 | 1 | 1
  Asian | 0 | 2 | 2
  Black/African American | 3 | 6 | 9
  Not reported | 1 | 0 | 1
  Unknown/other | 8 | 9 | 17
  White | 30 | 28 | 58
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 28.6 [24.8 to 32.7] | 30.6 [24.9 to 35.9] | 28.9 [24.8 to 34.7]
Past Medical History: Malignancy [Count of Participants; unit: Participants] | 8 | 10 | 18
Past Medical History: Coronary Artery Disease [Count of Participants; unit: Participants] | 10 | 8 | 18
Past Medical History: Congestive Heart Failure [Count of Participants; unit: Participants] | 9 | 13 | 22
Past Medical History: Liver Disease [Count of Participants; unit: Participants] | 0 | 6 | 6
Chronic Kidney Disease [Count of Participants; unit: Participants] — Participants were staged using the KDIGO (Kidney disease - improving global outcomes) classification of the stages of chronic kidney disease, which uses the clinically observed glomerular filtration rate (GFR) to classify patients. A decreased GFR indicates a higher "stage" of KDIGO and thus corresponds to a worse outcome [A patient with stage 4 is sicker than a patient with stage 2].
  Participants
    No Kidney Disease | 34 | 38 | 72
    Stage 2 | 1 | 1 | 2
    Stage 3a | 2 | 1 | 3
    Stage 3b | 2 | 1 | 3
    Stage 4 | 0 | 2 | 2
    Unknown/not reported | 3 | 3 | 6
Source of Sepsis [Count of Participants; unit: Participants]
  Endocarditis | 0 | 2 | 2
  Infection of unknown source | 3 | 3 | 6
  Intra-abdominal infection | 10 | 9 | 19
  Other | 6 | 5 | 11
  Pneumonia | 7 | 9 | 16
  Skin or soft tissue infection | 4 | 2 | 6
  Urinary tract infection | 12 | 16 | 28
Volume of intravenous fluids prior to study drug [Median (Inter-Quartile Range); unit: mL] | 2000 [1361.5 to 3500.0] | 1819.0 [907.8 to 3214.5] | 1972.5 [1138.8 to 3500.0]
Baseline cardiovascular component of the total SOFA score [Median (Inter-Quartile Range); unit: units on a scale] — Score on a scale that ranges from 0-24, with 24 being the worst outcome.
  units on a scale | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
Time from vasopressor initiation to first study drug [Median (Inter-Quartile Range); unit: Hours] | 12.8 [8.3 to 24.0] | 14.4 [8.2 to 23.7] | 14.1 [8.2 to 24.2]
Time from informed consent to first study drug [Median (Inter-Quartile Range); unit: Hours] | 1.6 [1.4 to 2.2] | 1.6 [1.3 to 1.9] | 1.6 [1.3 to 2.0]
Mechanically ventilated [Count of Participants; unit: Participants] | 27 | 27 | 54
Lactate [Median (Inter-Quartile Range); unit: mmol/L] | 2.9 [2.3 to 4.4] | 3.1 [2.5 to 4.7] | 2.9 [2.4 to 4.7]
30-day predicted survival [Count of Participants; unit: Participants]
  High likelihood | 10 | 8 | 18
  Uncertain | 29 | 37 | 66
  Low likelihood | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Kidney Injury Biomarker
Description: Change in creatinine over time
Time Frame: Enrollment to 72-hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 42 | 46
mg/dL | 2.24 (1.50) | 2.79 (1.91)
Statistical Analysis 1: Comparison: Thiamine vs Placebo; Test type: Other; p = 0.07, Mixed Models Analysis — Mixed model controlling for repeated measures within patients used to get a mean difference in creatinine between the thiamine and placebo groups at 72 hours. Missing creatinine imputed using a penalty (20pc increase) as described in SAP; P-value is for the comparison at 72 hours from the mixed model (i.e, not a global p-value); Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-1.18 to 0.04]

2. Secondary Outcome: Number of Participants Receiving Renal Replacement Therapy
Description: Number of participants who received renal replacement therapy in thiamine and placebo groups.
Time Frame: From date of enrollment until discharge from the intensive care unit (ICU) or date of death, whichever comes first, up to 60 days after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 42 | 46
Participants | 6 | 10
Statistical Analysis 1: Comparison: Thiamine vs Placebo; Test type: Other; p = 0.34, Regression, Logistic — P-value from odds ratio from logistic regression model controlling for site, with outcome of receiving renal replacement therapy; Odds Ratio (OR) = 0.58, 95% CI 2-sided [0.18 to 1.74]

3. Secondary Outcome: ICU Free Days
Description: Days alive and free of the ICU through day 28
Time Frame: From date of enrollment until 28 days after enrollment
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 42 | 46
days | 22.5 [0.0 to 25.0] | 0.0 [0.0 to 23.0]
Statistical Analysis 1: Comparison: Thiamine vs Placebo; Test type: Other; p = 0.002, Quantile regression — P-value from quantile regression model controlling for site; Median Difference (Final Values) = 22.0, 95% CI 2-sided [7.4 to 36.6]

4. Secondary Outcome: In-hospital Mortality
Description: Length of hospital stay truncated at 60 days
Time Frame: From date of enrollment until discharge from the hospital or date of death, whichever comes first, up to 60 days after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 42 | 46
Participants | 15 | 25
Statistical Analysis 1: Comparison: Thiamine vs Placebo; Test type: Other; p = 0.14, Regression, Cox — P-value from Cox proportional hazards model adjusting for site; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.32 to 1.18]

5. Secondary Outcome: Number of Participants Experiences Acute Renal Failure
Description: Acute renal failure as defined by the KDIGO (Kidney Disease Improving Global Outcomes) AKI (Acute Kidney Injury) criteria. In brief, a patient can meet these criteria if their serum creatinine increases (for example, serum creatinine increases to 1.5x or higher of baseline serum creatinine, or if it crosses 4mg/dL), or if renal replacement therapy is initiated, or if urine output decreases (for example, <0.5ml/kg/hour for 6-12 hours) or if patient becomes anuric (no urine production).
Time Frame: From date of enrollment until day of discharge from the index ICU admission or date of death, whichever comes first up until 60 days post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 42 | 46
Participants | 23 | 34
Statistical Analysis 1: Comparison: Thiamine vs Placebo; Test type: Other; p = 0.07, Regression, Logistic — P-value from logistic regression model controlling for site; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.17 to 1.06]

6. Secondary Outcome: Change in Lactate Level
Description: Change in lactate level between enrollment and 72 hours after enrollment
Time Frame: From time of enrollment until 72 hours after enrollment
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 42 | 46
mmol/L | 1.65 [1.10 to 2.80] | 1.95 [1.40 to 2.30]
Statistical Analysis 1: Comparison: Thiamine vs Placebo; Test type: Other; p = 0.79, Mixed Models Analysis — Mixed model controlling for repeated measures within patients used to get a mean difference in lactate between the thiamine and placebo groups at 72 hours. Missing lactate imputed using a penalty (20pc increase) as described in SAP; P-value is for the comparison at 72 hours from the mixed model (i.e, not a global p-value); Mean Difference (Final Values) = 0.96, 95% CI 2-sided [0.71 to 1.30]

7. Secondary Outcome: Number of Participants With Delirium on Day 3
Description: Number of Participants with Delirium on Day 3 after enrollment
Time Frame: Day 3 after enrollment
Population: Excludes 8 and 4 patients in intervention and placebo groups with delirium status "unable to assess"
Measure: Count of Participants; unit: Participants
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 34 | 42
Participants | 25 | 30

8. Secondary Outcome: Change in the Sequential Organ Failure Assessment Score
Description: Change in Sequential Organ Failure Assessment Score (SOFA) score between enrollment and 72 hours after enrollment. SOFA scores are reported on a scale between 0-24, with 0 representing best outcome and 24 representing worst outcome.
Time Frame: Time of enrollment until 72 hours after enrollment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 42 | 46
units on a scale | 8.09 (5.60) | 9.61 (5.96)
Statistical Analysis 1: Comparison: Thiamine vs Placebo; Test type: Other; p = 0.16, Mixed Models Analysis — Mixed model controlling for repeated measures within patients used to get a mean difference in SOFA scores between the thiamine and placebo groups at 72 hours. Missing SOFA imputed using a penalty (20pc increase) as described in SAP; P-value is for the comparison at 72 hours from the mixed model (i.e, not a global p-value); Mean Difference (Final Values) = -1.53, 95% CI 2-sided [-3.63 to 0.58]

9. Secondary Outcome: Novel Biomarkers of Renal Injury
Description: KIM-1, NGAL, Cystatin-C at 24-hours after enrollment
Time Frame: 24 hours after enrollment
Population: A total of 32 patients in thiamine and 37 patients in placebo had biomarkers available at both 0 hours and 24 hours and thus contributed to the model estimates
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Thiamine | Placebo
Number analyzed (Participants) | 32 | 37
pg/mL
  KIM-1 | 763.1 [454.8 to 1504.8] | 793.9 [350.6 to 1548.8]
  NGAL | 1067898.2 [501797.2 to 1528804.4] | 1558285.0 [966335.0 to 3235305.6]
  Cystatin | 1689158.2 [1238353.1 to 2677488.6] | 2183175.4 [1614104.4 to 2819738.6]

ADVERSE EVENTS:
Time Frame: From enrollment to time of discharge, an average of 2 weeks.
Description: As detailed in the clinical trial protocol.
Arm/Group | Thiamine | Placebo
All-Cause Mortality (participants affected / at risk) | 15/42 | 25/46
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/46
Other Adverse Events (participants affected / at risk) | 0/42 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT03550794/Prot_001.pdf
  • Statistical Analysis Plan (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT03550794/SAP_000.pdf